CLINICAL TRIAL: NCT01860586
Title: A Prospective Pilot Study Evaluating the Effect of Intravitreal Injection of Bevacizumab on Recurrent Retinal Detachment Due to Proliferative Vitreoretinopathy
Brief Title: Eye Injections of Bevacizumab for Lowering Risk of Scar Tissue in the Retina and Repeated Retinal Detachment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jason Hsu, MD, Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HsuPVR13; MARPVR2013 (Other: Mid Atlantic Retina)
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Retinal Detachment; Vitreoretinopathy Proliferative
Keywords: pvr; rd; Proliferative Vitreoretinopathy; retinal detachment; detachment
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Outcomes were compared to a retrospective, historical control group.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab will be injected into the study eye at end of retinal detachment (rd) surgery and monthly for the following 3 months (total of 4 intravitreal bevacizumab injections)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (1.25mg/0.05mL) will be injected into the study eye, at the end of the surgical repair of the retinal detachment and at Month 1, 2 and 3.
  Other Names: Avastin; Intrasilicone oil intravitreal injection

SUMMARY:
The purpose of this study is to examine the effects of a drug called bevacizumab (Avastin) on the rates of recurrent retinal detachment and scar tissue formation.

DETAILED DESCRIPTION:
Proliferative vitreoretinopathy (PVR) remains the most significant obstacle to successful retinal detachment (RD) repair, accounting for up to 75% of all primary surgical failures. Characterized by the proliferation of cells on the preretinal or subretinal surface, PVR ultimately leads to contraction, foreshortening, and ultimately recurrent detachment of the retina. Several PVR risk factors have been identified, including pre-existing uveitis, large retinal tears, multiple retinal breaks, detachments involving greater than two quadrants of the retina, vitreous hemorrhage, and choroidal detachment. Given the absence of a proven medical therapy for PVR and prior studies establishing VEGF as a potential therapeutic target, further clinical evaluation is warranted. Herein, we report outcomes of a prospective, non-randomized, historical-control pilot study evaluating the effect of serial intrasilicone oil bevacizumab injections on outcomes of PVR-related RD repair.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Undergoing pars plana vitrectomy with or without scleral buckling for recurrent RD due to PVR with planned silicone oil instillation.

Exclusion Criteria:

* Prior anti-VEGF (vascular endothelial growth factor) injections within 3 months of retinal detachment surgery.
* Traction retinal detachment due to proliferative diabetic retinopathy.
* Inability to flatten retina completely intraoperatively
* Known allergy or contraindication to intravitreal bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — WillsEye Hospital
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Bevacizumab will be injected into the study eye at end of retinal detachment (rd) surgery and monthly for the following 3 months (total of 4 intravitreal bevacizumab injections)
  Bevacizumab: .05 mL of Bevacizumab will be injected into the study eye, at the end of the surgical repair of the retinal detachment and at Month 1, 2 and 3.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Intravitreal Bevacizumab Injections on Rate of Recurrent Retinal Detachment (Increase or Decrease)
Description: This will be assessed by the frequency (occurences) of retinal detachments in patients that have intravitreal bevacizumab injections versus prior patients that did not have intravitreal bevacizumab injections.
Time Frame: up to 6 months
Population: Bevacizumab treated patients with recurrent retinal detachment
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab: Bevacizumab will be injected into the study eye at end of retinal detachment (rd) surgery and monthly for the following 3 months (total of 4 intravitreal bevacizumab injections)
  Bevacizumab: .005 mL of Bevacizumab will be injected into the study eye, at the end of the surgical repair of the retinal detachment and at Month 1, 2 and 3.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
Participants | 6

2. Secondary Outcome: The Effect of Intravitreal Bevacizumab Injections on the Development of Epiretinal Membranes (Increase or Decrease)
Description: To determine if intravitreal bevacizumab injections will increase or decrease the occurences (cases) of epiretinal membranes .
Time Frame: 6 months
Population: Number of patients treated with bevacizumab who developed epiretinal membrane
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
Participants | 7

3. Other Pre Specified Outcome: Intravitreal Bevacizumab Injections Impact on Visual Acuity Score (Change in Letters Read).
Description: Increase or decrease in amount of letters read after intravitreal bevacizumab injections versus control patient that did not receive injections of intravitreal bevacizumab.
Time Frame: 6 months
Population: Final logMAR visual acuity of patients treated with bevacizumab
Measure: Mean (Standard Deviation); unit: logMAR visual acuity
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
logMAR visual acuity | 1.43 (0.70)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Systematic assessment via investigator examinations.
Arm/Group | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This pilot study has several limitations, including small sample size, its non-randomized nature, and use of historical controls for outcome comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes